CLINICAL TRIAL: NCT02942550
Title: Methylnaltrexone as a Method to imprOVE Platelet Inhibition of Ticagrelor in Morphine-treated Patients With ST-segMENT Elevation Myocardial Infarction: a Prospective, Single Blinded Randomized, Placebo-controlled Trial
Brief Title: Methylnaltrexone as a Method to Improve Ticagrelor Uptake in Morphine Treated STEMI Patients
Acronym: MOVEMENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jan van der Linden, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 880526
Record Dates: First submitted 2016-09-21; First posted 2016-10-24 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: STEMI; Morphine; Ticagrelor; Methylnaltrexone
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — methylnaltrexone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylnaltrexone (Active Comparator): Methylnaltrexone bromide (Relistor®). Single intravenous injection of 8 mg (0.4 ml solution) for patients weighing 38-61 kg or 12 mg (0.6 ml solution) patients weighing 62-114 kg).
  Interventions: Drug: Methylnaltrexone bromide (Relistor®).
- Placebo (Placebo Comparator): Sodium Chloride, 9mg /mL ingle intravenous injection of 0.4 mL solution for patients weighing 38-61 kg or 0.6 mL solution patients weighing 62-114 kg).
  Interventions: Drug: Sodium Chloride 9mg/mL

INTERVENTIONS:
Drug: Methylnaltrexone bromide (Relistor®).
  Arms: Methylnaltrexone
Drug: Sodium Chloride 9mg/mL
  Arms: Placebo

SUMMARY:
This study will examine the impact of the peripheral opioid antagonist methylnaltrexone on the onset of effect of ticagrelor in morphine treated patients with ST elevation myocardial infarction (STEMI). Half of the participants will receive methylnaltrexone, while the other half will receive placebo.

DETAILED DESCRIPTION:
The rate of drug absorption in the gastro-intestinal tract is often determined by the rate of gastric emptying. Morphine treatment, which is frequently given in order to relieve pain in patients with STEMI, is known to delay gastric emptying, and has indeed emerged as a predictor of delayed/poor antiplatelet response in patients receiving oral prasugrel or ticagrelor.

In recent years, morphine has been found to delay the onset of oral P2Y12-inhibitors. To counteract this, the investigators hypothesized that an opioid antagonist may be used. The opioid antagonist naloxone has previously been shown to reduce the morphine induced delay in gastric emptying However, naloxone crosses the blood-brain barrier (BBB) and reduces the pain relieving effects of morphine. In contrast, the morphine antagonist methylnaltrexone has a reduced passage over the BBB and acts primarily as a peripheral morphine antagonist without affecting the morphine-mediated central analgesic effects.

The aim of the planned study is to evaluate whether methylnaltrexone bromide may reduce the morphine induced delay in onset of platelet inhibition after a loading dose of 180 mg ticagrelor in morphine treated patients with STEMI undergoing primary percutaneous coronary intervention (PCI), where a rapid and adequate platelet inhibition after the administration of ticagrelor is crucial. As morphine is an inclusion criterion, all patients included in the study will be on morphine treatment. Thus, morphine treatment is not an intervention to be administered as part of the protocol. Stratification according to inferior and anterior/lateral STEMI will be perform to avoid imbalance in the location of myocardial infarction between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of STEMI
* Administration of a 180 mg loading dose ticagrelor
* Analgesic treatment with intravenous morphine pre-PCI

Exclusion Criteria:

* Cardiac arrest
* Body weight > 114kg
* Vomiting after intake of ticagrelor loading dose
* Use of Naloxone before inclusion or during sampling period
* Inability to understand study outline and instructions
* Methylnaltrexone bromide contraindication
* Age <18 years; 8) Women in fertile age
* Administration of ticagrelor during the week before inclusion
* Treatment with Cangrexal
* Ongoing long-term opioid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
High on-treatment platelet reactivity (HPR) | Two hours after the injection of either active drug or placebo
  HPR defined as platelet reactivity index (PRI) ≥50% using VASP analysis
Number of participants with serious adverse events | Within 48 hours after drug administration
  Serious AE is any untoward medical occurrence that at any dose:
  * Results in death.
  * Is life-threatening at the time of the event.
  * Requires inpatient hospitalization.
  * Requires prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Is a congenital anomaly/birth defect.

SECONDARY OUTCOMES:
High on-treatment platelet reactivity | One hour after the injection of either active drug or placebo
Difference in ticagrelor and AR-C124910XX concentrations | One and two hours after the injection of either active drug or placebo
Change in patient pain according to visual analog scale | One and two hours after the injection of either active drug or placebo
Difference in ticagrelor and AR-C124910XX concentrations between patients with inferior STEMI and patients with anterior/lateral STEMI. | One and two hours after the injection of either active drug or placebo
Difference in high on-treatment platelet reactivity (HPR) between patients with inferior STEMI and patients with anterior/lateral STEMI. | One and two hours after the injection of either active drug or placebo
  HPR defined as platelet reactivity index (PRI) ≥50% using VASP analysis

CONTACTS AND LOCATIONS:
Overall Officials: Per Tornvall, MD, PhD, Principal Investigator — Karolinska Institutet; Ulf Jensen, MD, PhD, Principal Investigator — Karolinska Institutet; Nawzad Saleh, MD, PhD, Principal Investigator — Karolinska Institutet; Loghman Henareh, MD; PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Södersjukhuset (Stockholm South General Hospital), Stockholm

IPD SHARING:
Plan to Share IPD: No
Data will only be published on a group level.

REFERENCES:
- [Derived] Holm M, Tornvall P, Henareh L, Jensen U, Golster N, Alstrom P, Santos-Pardo I, Witt N, Fedchenko N, Venetsanos D, Beck O, van der Linden J. The MOVEMENT Trial. J Am Heart Assoc. 2019 Jan 22;8(2):e010152. doi: 10.1161/JAHA.118.010152. PMID 30636504